CLINICAL TRIAL: NCT05014347
Title: Patient Reported Experience Measure in Endoscopic Ultrasonography: the PREUS Study
Brief Title: Patient Reported Experience in Endoscopic Ultrasound
Acronym: PREUS
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Paolo Giorgio Arcidiacono, MD, MD FASGE Associate Professor of Gastroenterology, Vita-Salute San Raffaele University; Head Pancreatico/Biliary Endoscopy & Endosonography Division Pancreas Translational & Clinical Research Center San Raffaele Scientific Institute, Milan,Italy, IRCCS San Raffaele
Other Study IDs: PREUS
Record Dates: First submitted 2021-08-13; First posted 2021-08-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Diseases; Bile Duct Diseases
Keywords: patient reported experience measures; endoscopic ultrasonography; pancreatic; questionnaire
MeSH Terms: conditions — Pancreatic Diseases; Bile Duct Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Health Care Professionals: Health Care Professionals (HCP) working in PancreatoBiliary Endoscopy and EUS Division of IRCCS San Raffaele (both endoscopists and nurses)
- "Expert" patients: a set of at least 30 outpatients undergoing EUS, who already underwent this procedure at least once
- Patients: 100 consecutive patients undergoing EUS

SUMMARY:
The evaluation of the patient's experience is becoming increasingly important as a better patient experience can improve the quality of the delivered health service. Patient-reported experience measures (PREMs) are self-reported assessment tools provided by patients about their experience during any health event. There are few PREMs's instruments in the field of gastrointestinal endoscopy, and none is specific for Endoscopic Ultrasound (EUS). The aim of this study is to develop a questionnaire to evaluate the experience of patients undergoing EUS, identifying and prioritizing the factors related to the patient's experience. In order of it, expected results are developing a valid tool of question to value patients experience during EUS and, for ranking, it is iphotized that will be more correlation with patients's and nurses's answer that clinicians's one. In literature is described that nurse's view and patient's view are more similar especially in those aspects concerning empatics and psychological aspects.

DETAILED DESCRIPTION:
The study will consist of several phases: 1) Tool creation: a "patient reported measure of EUS" (PREUS) questionnaire will be created based on literature review; 2) Face and Content Validity: The PREUS tool will be submitted to 7 experts in the field (physicians, nurses, psychologist, communication expert, patients' advocacy representative) for a two-round evaluation and to "expert" patients who had already undergone EUS at least once. Content Validity Index (CVI) will be calculated and questions with a CVI < 0.70 will be excluded; 3) Questionnaire Creation: Based on the results of phase 2, a modified "PREUS" tool will be then evaluated by ranking the relevance of the identified questions in the previous phase (from 0 to 10) by 50 outpatients undergoing EUS and Cronbach's alpha will be calculated to determine reliability; 4) Ranking: tool of phase 3 will be also evaluated by 6 physicians and 13 nurses working in IRCCS Ospedale San Raffaele endoscopy Unit to measure the agreement between patients and health care professionals (HCPs) by the Spearman-Brown coefficients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Outpatients undergoing EUS in I.R.C.C.S. San Raffaele Hospital (Milan, Lombardy, Italy);
* Written informed consent signed

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Outpatients undergoing EUS in I.R.C.C.S. San Raffaele Hospital (Milan, Lombardy, Italy); HCP involved with EUS in I.R.C.C.S S. Raffaele Hospital (OSR).
Sampling Method: Non-Probability Sample
Enrollment: 171 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
developing questionnaire | 9 months
  develop a questionnaire for Patient Reported Experience Measures during Endoscopic Ultrasound. In the first step it will be used a continuos Likert scale from 1 to 10 to analyse Content Validity Index, in the second step it will be used a score from 1 to 5 (1 = poor; 3 = good; 5 = excellent experience)

SECONDARY OUTCOMES:
ranking | 9 months
  identify aspects of care that are most relevant both for patients undergoing EUS and HCPs involved in this procedure on a continuous Likert scale from 1 to 10 (1 = less important; 5 = relatively important; 10 = more important).

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriele Capurso, Milan, Italy